CLINICAL TRIAL: NCT02149602
Title: A Phase II Study of Parotid-gland Sparing Intensity-modulated Radiotherapy in Patients With Midline Tumour of the Head and Neck
Brief Title: A Phase II Study of Parotid-gland Sparing IMRT in Patients With Midline Tumour of the Head and Neck
Acronym: PARSPORT-II
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 2588
Record Dates: First submitted 2014-05-26; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Oropharyngeal Squamous Cell Cancer; Hypopharyngeal Squamous Cell Cancer
Keywords: involvement of bilateral parapharyngeal spaces
MeSH Terms: interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- oropharyngeal and hypopharyngeal HNSCC: Intensity Modulated Radiotherapy HPV positive and HPV negative
  Interventions: Radiation: Intensity modulated radiotherapy

INTERVENTIONS:
Radiation: Intensity modulated radiotherapy — Bilateral superficial lobe parotid sparing intensity modulated radiotherapy

SUMMARY:
This study is a phase II trial designed to test the feasibility of delivering IMRT to head and neck cancer patients with tumours arising in the midline (oropharynx and hypopharynx), and to assess possible improvement in reducing the incidence of xerostomia with bilateral superficial lobe parotid sparing IMRT.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed locally advanced HNSCC arising from the oropharynx or hypopharynx with high risk of bilateral parapharyngeal space involvement

Exclusion Criteria:

* Patients <18 years old or with a previous malignancy other than non-melanomatous skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Midline pharyngeal squamous cell cancers (excluding nasopharyngeal cancers)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2005-07; Primary Completion 2011-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
The proportion of patients reporting grade 2 or more xerostomia using subjective measure on the LENTSOMA late toxicity scoring scale one year after treatment. | 12 months

SECONDARY OUTCOMES:
Acute radiation toxicity | 0-3 months
Late radiation toxicity | 3-24 months
Survival outcomes for entire cohort and according to HPV status where available : Local control, Loco regional control, Loco-regional progression-free survival (LRPFS), Disease free survival, Overall survival. | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Nutting, FRCR, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Head and Neck Unit, Royal Marsden Hospital, London, United Kingdom